CLINICAL TRIAL: NCT05285124
Title: Effect and Mechanism of HD-tDCS Combined With Circadian Rhythm Remodeling on Consciousness Recovery in Patients With Chronic Disorder of Consciousness
Brief Title: HD-tDCS Combined With Circadian Rhythm Reconstruction and Micro Expression Changes on Consciousness Recovery in Patients With Chronic Disturbance of Consciousness
Acronym: HD-tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Sleep and stimulation
Record Dates: First submitted 2021-05-17; First posted 2022-03-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-04

CONDITIONS: Disorder of Consciousness
Keywords: disorder of consciousness; Circadian rhythm; HD-tDCS
MeSH Terms: conditions — Consciousness Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- tDCS and melatonin intervention (Experimental): In real tDCS, the current was increased to 2 mA from the onset of stimulation and applied for 20 minutes. Participants were given a 3-mg fast-release oral dose of melatonin.
  Interventions: Drug: Melatonin; Other: HD-tDCS
- tDCS intervention (Experimental): In real tDCS, the current was increased to 2 mA from the onset of stimulation and applied for 20 minutes.
  Interventions: Other: Placebo; Other: HD-tDCS
- Melatonin intervention (Experimental): Participants were given a 3-mg fast-release oral dose of melatonin.
  Interventions: Drug: Melatonin
- Control (Placebo Comparator): Patients were treated with the placebo and sham-tDCS.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Participants assigned to the melatonin group were given a 3-mg fast-release oral dose of melatonin administered at approximately 21:00
  Arms: Melatonin intervention; tDCS and melatonin intervention
Other: Placebo — Participants in this group were treated according to a protocol identical to those receiving active medication at approximately 21:00. For the sham tDCS groups, the same stimulation parameters were employed, except that the stimulator had a built-in placebo mode; when it was activated, two ramp fade-in/fade-out periods in the beginning and the end of sham stimulation mimicked the somatosensory artifact of real tDCS
  Arms: Control; tDCS intervention
Other: HD-tDCS — Direct current was applied using a battery-driven constant-current stimulator through saline-soaked surface sponge electrodes (7cm×5cm) with the anode placed over the left DLPFC (F3 according to the 10-20 international EEG system) and the reference cathode placed over the right supraorbital region (Fp2). During real tDCS, the current was increased to 2 mA from the onset of stimulation and applied for 20 minutes
  Arms: tDCS and melatonin intervention; tDCS intervention

SUMMARY:
The circadian rhythm characteristics of sleep cycle and neuroendocrine in patients with chronic disorder of consciousness show different degrees of disorder, and the relationship between this disorder and consciousness level is unclear.The researchers used HD-tDCS to treat patients with chronic disturbance of consciousness who intervened in circadian rhythm, and used a variety of methods such as EEG, fMRI, protein metabolism, ERP and micro-expression to explore the mechanism of improving the state of consciousness of HD-DCS and the relationship between circadian rhythm and patients' consciousness level

DETAILED DESCRIPTION:
The sleep status (> 24 hours) of patients with chronic disturbance of consciousness was recorded with the revised coma recovery scale revised (CRS-R) and Polysomnography (PSG). The sleep cycle of patients with chronic disturbance of consciousness was judged by the open and close eyes cycle and EEG.

Patients with circadian rhythm treated with or without blue light stimulation and melatonin were treated with HD-tDCS. EEG, fMRI, protein metabolism, ERP and micro expression data were recorded before and after treatment.Explore the mechanism of improving the state of consciousness of HD-DCS and the relationship between circadian rhythm and patients' consciousness level

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of disorder of consciousness
* Stable vital signs
* Good coordination, less spontaneous activity
* No anti-epileptic and sedative drugs taken within prior 24 hours
* The family members volunteered and signed the informed consent

Exclusion Criteria:

* locked-in syndrome
* Diseases and factors that may affect the judgment of brain function, such as metabolic diseases, poisoning, shock, etc.
* There are contraindications to MRI scanning, such as the presence of metal implants in the body
* Contraindications treated by transcranial direct current stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Coma Recovery Scale-Revised (CRS-R) scale | Change from Baseline CRS-R at 14 days.
  The CRS-R is a tool used to characterise the level of consciousness consisting of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The values range from 0 to 23, with higher score indicating better outcome.
Electroencephalography (EEG) | Change from baseline EEG power spectral density at 14 days.
  Delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz) and beta (12-30 Hz). An increase of delta and theta activity usually reflects encephalopathy and/or structural lesions, interpreted as poor outcome predictor of DOC .The power of α and β is related to the chance of recovery.
Sleep parameters | Change from baseline sleep patterns at 14 days.
  Changes in in sleep/wake architecture assessed by polysomnography. Electrodes attached to the scalp near the frontal, central (top) and occipital (back) portions of the brain and provide a readout of different stages of sleep (N1, N2, N3, REM, and Wakefulness).
Resting state fMRI | Change from ReHo, ALFF, fALFF and functional connectivity at 14 days.
  Resting state fMRI reflects the brain activity occured in a resting or task-negative state. Regional (ReHo, ALFF, fALFF, etc.) and global parameters (functional connectivity, etc.) could be used in this study.
Micro-expression | At baseline.
  After listening to auditory stimulations, transient alterations may occur on the micro expression of the subjects. High-resolution video will be taken to capture each subject's facial micro-expressions while listening to the auditory materials.

SECONDARY OUTCOMES:
protein metabolism | Change from Baseline protein metabolism at 14 days.
  Changes of protein content in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, PhD, Study Director — The First Affiliated Hospital, Zhejiang University
Locations (1):
- First Affiliated Hospital,Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen X, Yu J, Zhu G, Wang J, Sun Y, Zhou J, Cai J, Meng F, Ling Y, Sun Y, Zhao J, He F, Cheng Q, Xu C, Gao J, Li J, Luo B. Efficacy of melatonin for prolonged disorders of consciousness: a double-blind, randomized clinical trial. BMC Med. 2024 Dec 3;22(1):576. doi: 10.1186/s12916-024-03793-2. PMID 39627786